CLINICAL TRIAL: NCT01374815
Title: The Online Advocate: Health Related Social Problems And Diet Quality Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Clement Bottino, Principal investigator, study coordinator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: X10-07-335
Record Dates: First submitted 2011-06-13; First posted 2011-06-16 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Children's Diet Quality; Health-related Social Problems
Keywords: Children's diet quality; Health-related social problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Online Advocate (Experimental)
  Interventions: Other: The Online Advocate

INTERVENTIONS:
Other: The Online Advocate — The Online Advocate is a Web-based social problems screening and referral tool developed at Children's Hospital.
Other: The Online Advocate — The Online Advocate is a Web-based screening and referral tool for health-related social problems

SUMMARY:
In this study, the investigators will be using The Online Advocate, a Web-based health-related social problems screening and referral tool, to explore the relationship between health-related social problems and children's diet quality among families with young children attending the Children's Hospital Primary Care Center. The Online Advocate consists of a 60-80 question screening survey for health-related social problems (such as food insecurity, employment and income, homelessness) and allows participants to select referrals for local health and social service agencies that might help them with the problems identified through the survey. Layered into The Online Advocate for this study is an adaptation of the Harvard Service Food Frequency Questionnaire (HSFFQ) that can assess children's diet quality. The investigators plan to recruit 350 parent/guardians of otherwise healthy children age 3-10 years who are presenting to the primary care center for routine well child care. Eligible parent/guardians will have the opportunity to take The Online Advocate (plus HSFFQ) on a laptop computer in the waiting area before seeing their pediatrician or healthcare provider. Participants will receive a small incentive for their time as well as written information on healthy nutrition and an age appropriate coloring book for the child. At one month, participants will be contacted by the study team by email or phone and asked follow up questions about the status of their health-related social problems identified through The Online Advocate and whether the referrals they received were helpful. Participants will receive a small incentive for their time, along with a reminder message promoting healthy nutrition for their child. At three months, participants will be contacted by the study team by email or phone and asked follow up questions about the status of their health-related social problems identified through The Online Advocate and whether the referrals they received were helpful. They will also re-take the adapted HSFFQ. Participants will receive another small incentive for their time. Participants will also have the opportunity to re-take The Online Advocate at three months, though this is optional. The investigators believe this pilot study will provide foundational knowledge about the intersection between health-related social problems and children's diet quality and may inform future research studies and interventions.

Our Study Aims are:

1. To use The Online Advocate to evaluate the association between health-related social problems and diet quality in children in a cross-sectional sample.
2. To evaluate the relationship between resolution of health-related social problems using The Online Advocate and change in diet quality in children over a 3 month period.

Our Study Hypotheses are:

1. A greater number of health-related social problems per family will be associated with poorer diet quality in children at baseline.
2. After 3 months, families demonstrating resolution of one or more health-related social problems addressed with The Online Advocate will demonstrate greater improvement in diet quality in children.

ELIGIBILITY:
Inclusion Criteria:

* Child age 3 to 10 years
* Child lives with parent/guardian at least 5 days per week
* Parent/guardian must be able to speak and read in English

Exclusion Criteria:

* Child with major, active chronic medical illness (e.g., cancer) or use of prescription medication (e.g., oral steroids) that might influence diet quality
* Prior use of The Online Advocate
* Prior study participation
* Child is first degree relative (e.g., sibling) of current or prior study participant or a family member with lesser degree of relatedness or non-relative who lives in the same household as a current or prior study participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Diet quality | 3 months
  Diet quality will be assessed using the HEI-2005, Healthy Eating Index, applied to the nutritional data collected using the HSFFQ survey. HEI-2005 provides an overall score (scale 0 to 100) and was developed by the USDA Center for Nutrition Policy and Promotion to assess compliance with dietary guidelines.

SECONDARY OUTCOMES:
Physical activity | 3 months
  Physical activity will be assessed using the NHANES survey.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne E Cox, MD, Principal Investigator — Boston Children's Hospital; Clement J Bottino, MD, Study Director — Boston Children's Hospital; Erinn T Rhodes, MD, MPH, Principal Investigator — Boston Children's Hospital; Eric W Fleegler, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bottino CJ, Fleegler EW, Cox JE, Rhodes ET. The Relationship Between Housing Instability and Poor Diet Quality Among Urban Families. Acad Pediatr. 2019 Nov-Dec;19(8):891-898. doi: 10.1016/j.acap.2019.04.004. Epub 2019 Apr 13. PMID 30986548